CLINICAL TRIAL: NCT04976088
Title: Randomized, Double Blind, Parallel-groups, Non-inferiority Versus Flector® and Superiority Versus Placebo, Phase III Clinical Trial With Diclofenac Sodium 140 mg Medicated Plaster in Patients With Impact Injuries of the Limbs
Brief Title: Clinical Trial With Diclofenac Sodium Medicated Plaster in Patients With Impact Injuries of the Limbs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EQI7_16_02
Record Dates: First submitted 2020-03-02; First posted 2021-07-26 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Trauma Injury; Inflammation
Keywords: traumatic
MeSH Terms: conditions — Accidental Injuries; Inflammation | interventions — Diclofenac; diclofenac hydroxyethylpyrrolidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A Test (Experimental): Test product: treated once a day (morning) with the medicated plaster containing 140 mg Diclofenac Sodium for seven days Diclofenac Sodium 140 mg medicated plaster
  Interventions: Drug: Diclofenac Sodium 140 mg medicated plaster
- Group B Reference (Active Comparator): Reference product: treated once a day (morning) with the medicated plaster containing DIEP 180 mg, Flector® for seven days Diclofenac epolamine (DIEP) 180 mg medicated plaster, Flector®
  Interventions: Drug: Diclofenac epolamine (DIEP) 180mg medicated plaster, Flector
- Group C Placebo (Placebo Comparator): Placebo: treated once a day (morning) with the placebo plaster for seven days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac Sodium 140 mg medicated plaster — Test product: Diclofenac Sodium 140 mg medicated plaster, topical application once a day
  Other Names: EQI7
  Arms: Group A Test
Drug: Diclofenac epolamine (DIEP) 180mg medicated plaster, Flector — Reference product: Active-comparator, Diclofenac epolamine (DIEP) 180 mg medicated plaster, Flector®, topical application once a day
  Other Names: Flector
  Arms: Group B Reference
Drug: Placebo — Placebo: Placebo plaster, topical application once a day.
  Other Names: Placebo plaster
  Arms: Group C Placebo

SUMMARY:
Phase III, multinational, multicentre, randomized, prospective, double blind, parallel groups, placebo-controlled study to evaluate the analgesic effects of Test Diclofenac Sodium 140mg medicated plaster, Reference DIEP 180 mg medicated plaster, Flector® and Placebo plaster in patients with painful and phlogistic disease due to acute traumatic events of the limbs.

DETAILED DESCRIPTION:
This will be a Phase III, multinational, multicentre, randomized, prospective, double blind, parallel groups, placebo-controlled study to evaluate the analgesic effects of Test Diclofenac Sodium 140mg medicated plaster (once a day), Reference DIEP 180 mg medicated plaster, Flector® (once a day) and Placebo plaster once a day (i.e. the placebo arm) in patients with painful and phlogistic (inflammatory response) disease due to acute traumatic events (injury/contusion) of the limbs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age range 18-65 years (included);
2. Patient with painful and phlogistic (inflammatory response) disease due to acute traumatic events (injury/contusion) of the limbs;
3. Patient with pain at rest in only one limb surface area affected by injury/contusion;
4. Written informed consent to participate in the study obtained according to GCP;
5. Patients able to comprehend the full nature and the purpose of the study, including possible risks and side effects, and able to cooperate with the Investigator and to comply with the requirements of the entire study (including ability to attend all the planned study visits according to the time limits), based on Investigator's judgement;
6. Good general health as determined by the Investigator based on medical history and physical examination;
7. Female of child-bearing potential (i.e. not in menopausal status from at least one year or permanently sterilized) must have a negative urine pregnancy test prior the first IMP administration;
8. Presence of pain at rest in the injured area, defined by patient with a VAS ≥40 mm and ≤80 mm at Visit 1 on a 100 mm VAS

Exclusion Criteria:

1. Patient with a chronic painful or phlogistic disease (from more than three months);
2. Patient with painful or phlogistic disease arising from fractures or severe trauma events;
3. Pregnancy or lactation period throughout the whole study duration;
4. If female and of child-bearing potential, patient not using a highly effective method of birth control. Highly effective birth control methods include: combined hormonal contraception (containing estrogen and progestogen) associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence*;
5. Presence of concurrent skin disorders or open wounds in the area to be treated;
6. History of alcohol or drug abuse;
7. History of allergy or hypersensitivity or intolerance to diclofenac and/or to active or inactive excipients of formulation;
8. Known hypersensitivity to non-steroidal anti-inflammatory drugs and to paracetamol;
9. Use of non-steroid anti-inflammatory drugs and analgesics in the week before Visit 1 (with the exception of paracetamol, which should not be taken in the previous 8 hours), oral corticosteroids within 2 weeks or intravenous corticosteroids within 4 weeks before Visit 1. Chronic intake of small doses of acetylsalicylic acid (≤ 162 mg/day) taken for at least 30 days prior to the first dose of study medication for non-analgesic reasons may be continued (with no change on dosage) for the duration of the study;
10. Any other treatment or medication for the same or other indications that, according to its pharmacological properties and in the opinion of the Investigator, can alter the perception of pain (e.g. heparinoids or other anticoagulant agents, opioids, psychotropic agents, anti H1 agents or analgesics like glucocorticosteroids, etc.) in the week before Visit 1;
11. Any other concomitant treatment (e.g. cosmetics, ointments at the treated area) or medication that cannot be interrupted and interferes with the conduct of the trial;
12. History of active or suspected esophageal, gastric, pyloric channel, or duodenal ulceration or bleeding within 30 days before Visit 1;
13. History of uncontrolled chronic or acute concomitant disease (e.g. cardiac dysfunction, liver dysfunction, hemorrhagic diathesis, …) which, in the Investigator's opinion, would contraindicate study participation or confound interpretation of the results;
14. Known malignant diseases in the last 5 years;
15. Pre-treatment of the traumatic event (injury/contusion) target of this study. Previous cooling (with ice, cooling spray) is authorized prior to Visit 1 (but not in the three hours preceding Visit 1);
16. Anticipated poor compliance by the patient;
17. Previous participation in this clinical trial;
18. Any relevant surgical treatment during the previous 2 months or planned during the trial;
19. Patient with a history of serious psychiatric disorders;
20. Participation in any other clinical study within 30 days prior to Visit 1. *Note: According to 4.1 paragraph "Birth control methods which may be considered as highly effective" of the CTFG/Recommendations related to contraception and pregnancy testing in clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2018-10-27 (Actual); Study Completion 2018-10-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in VAS score (Visual Analogue Scale from 0 to 100 mm, where the left extreme means "No pain = 0" while the right extreme means "Worst Pain Imaginable = 100") for pain at rest at 72 ± 2 hours (Day 4) after treatment start. | 72 hours
  Non-inferior efficacy of Test (once a day) over Reference (once a day) in reduction of pain after 3 days post-Baseline (72± 2 hours, Day 4), and superior efficacy of Test and Reference to Placebo (once a day) in improving pain at rest at 72 ± 2 hours (Day 4) after Baseline in patients with painful and phlogistic disease due to acute traumatic events of the limbs. A 100-mm Visual Analogue Scale (VAS) will be used for the assessment of pain at rest, from 0 to 100, where "No pain = 0" while "Worst Pain Imaginable = 100".

SECONDARY OUTCOMES:
Area under the curve (AUC) for pain at rest at Day 4 and Day 8 (SPID0-4d and SPID0-8d) | Day 4 and Day 8
  To compare Test to Reference and Placebo with regard to pain relief (pain at rest and pain on movement) at Day 4 and Day8, assessed through the AUC (Area Under the Curve) of VAS measurements (Visual Analogue Scale from 0 to 100 mm, where the left extreme means "No pain = 0" while the right extreme means "Worst Pain Imaginable = 100") at Day 4 and Day 8.
Change from baseline of VAS (Visual Analogue Scale 0-100 mm, where "No pain = 0" and "Worst Pain Imaginable = 100") for pain at rest at the other study time-points (including patients' home measurements), from Day 1 to Day 8. | Day 1, Day 2, Day 3, Day 4, Day 5,Day 6, Day 7, Day 8
  To compare efficacy of the Test product to Reference and Placebo with regard to pain relief (pain at rest and pain on movement) from Day 1 to Day 8.
Time to resolution of pain at rest, measured through VAS Scale (Visual Analogue Scale 0-100 mm, where "No pain = 0" and "Worst Pain Imaginable = 100") during from Baseline to Day 8. | From Day 1 until the date of resolution of pain at rest (maximum Day 8)
  To compare efficacy of Test in comparison to Reference and Placebo with regard to time to resolution of pain (pain at rest and pain on movement), measured with VAS score (Visual Analogue Scale 0-100 mm, where "No pain = 0" and "Worst Pain Imaginable = 100").
Change from baseline in VAS score (Visual Analogue Scale 0-100 mm, where "No pain = 0" and "Worst Pain Imaginable = 100") for pain on movement at 72 ± 2 hours (Day 4) and at 168 ± 2 hours (Day 8) after treatment start | Day 4 and Day 8
  To compare efficacy of Test to Reference and Placebo with regard to pain relief (pain on movement), measured with VAS score (Visual Analogue Scale 0-100 mm, where "No pain = 0" and "Worst Pain Imaginable = 100") at Day 4 and Day 8.
Proportion of responder patients (defined as a decrease ≥ 50% of baseline VAS (Visual Analogue Scale 0-100 mm, where "No pain = 0" and "Worst Pain Imaginable = 100") for pain at rest and on movement) at 72 ± 2 hours (Day 4) after treatment start | Day 4
  To compare efficacy of Test to Reference and Placebo with regard to proportion of responders to pain relief (pain at rest and pain on movement) at Day 4, considering a decrease as ≥ 50% of baseline VAS (Visual Analogue Scale 0-100 mm, where "No pain = 0" and "Worst Pain Imaginable = 100")
Proportion of patients that used rescue medication (paracetamol) from Baseline to Day 8 usign a patient diary | From Baseline to Day 8
  To compare the proportion of patients that used rescue medication from Baseline to Day 8 among the three treatment arms (Test, Refrence and Placebo) using a patient diary
Amount of tablets of rescue medication consumed from Baseline to Day 8, using a patient diary | From Baseline to Day 8
  To compare the amount of consumption of tablets of paracetamol among the three treatment arms (Test, Refrence and Placebo) using a patient diary
IMP adhesion, performed daily by patients and at Day 4 and Day 8 by the open staff member; following 5-point ordinal scale: 0:≥90% adhered; 1:≥75% to <90% adhered; 2:≥50% to <75% adhered; 3:<50% adhered but not detached; 4:Plaster detached | Day 1, Day 2, Day 3, Day 4, Day 5,Day 6, Day 7, Day 8
  To compare the adhesion of Test to Reference and Placebo in the site of application from Baseline to Day 8, 5-point ordinal scale: 0:≥90% adhered; 1:≥75% to <90% adhered; 2:≥50% to <75% adhered; 3:<50% adhered but not detached; 4:Plaster detached
Safety as change from baseline to Day 8 evaluated by physical examination using observation, palpitation, percussion, and auscultation | Day 1, Day 2, Day3, Day 4, Day 5,Day 6, Day 7, Day 8
  To compare Test with Reference and Placebo in patient safety as change from baseline to Day 8 using observation, palpitation, percussion, and auscultation
Safety as change from baseline to Day 8 evaluated by systolic blood pressure measured in mmHg | Day 1, Day 2, Day3, Day 4, Day 5,Day 6, Day 7, Day 8
  To compare Test with Reference and Placebo in systolic blood pressure, measured in mmHg, as change from baseline to Day 8
Safety as change from baseline to Day 8 evaluated by diastolic blood pressure measured in mmHg | Day 1, Day 2, Day3, Day 4, Day 5,Day 6, Day 7, Day 8
  To compare Test with Reference and Placebo in diastolic blood pressure, measured in mmHg, as change from baseline to Day 8
Safety as change from baseline to Day 8 evaluated by heart rate measured in bpm | Day 1, Day 2, Day3, Day 4, Day 5,Day 6, Day 7, Day 8
  To compare Test with Reference and Placebo in heart rate, measured in bpm, as change from baseline to Day 8
Safety as change from baseline to Day 8 evaluated by tracking the number of patient withdrawals | Day 1, Day 2, Day3, Day 4, Day 5,Day 6, Day 7, Day 8
  To compare Test with Reference and Placebo in patient safety as change from baseline to Day 8, tracking the number of withdrawals
Safety as change from baseline to Day 8 evaluated by tracking the number of adverse events | Day 1, Day 2, Day3, Day 4, Day 5,Day 6, Day 7, Day 8
  To compare Test with Reference and Placebo in patient safety as change from baseline to Day 8, tracking the number of adverse events
Local tolerability (erythema) at the IMP application site by Investigator at Day 1, Day 4 and Day 8 based on a 8-point categorical scale, where 0=no evidence of irritation and 7=strong reaction spreading beyond test site | Day 1, Day 4 and Day 8
  To compare Test with Reference and Placebo in relation to the level of irritation on the application site
Local tolerability (itching) at the IMP application site by Investigator at Day 1, Day 4 and Day 8 based on a 4-point categorical scale, where 0=absent and 3=severe | Day 1, Day 4 and Day 8
  To compare Test with Reference and Placebo in relation to the level of itching on the application site
Local tolerability (burning) at the IMP application site by Investigator at Day 1, Day 4 and Day 8 based on a 4-point categorical scale, where 0=absent and 3=severe | Day 1, Day 4 and Day 8
  To compare Test with Reference and Placebo in relation to the level of burning on the application site
Local tolerability (local pain) at the IMP application site by Investigator at Day 1, Day 4 and Day 8 based on a 4-point categorical scale, where 0=absent and 3=severe | Day 1, Day 4 and Day 8
  To compare Test with Reference and Placebo in relation to the level of local pain on the application site
Global assessment of local tolerability at IMP administration site by Investigator and patient according to the following score: 3=excellent; 2=good; 1=fair; 0=poor, assessed at Day 4 and Day 8. | Day 4 and Day 8
  To compare Test with Reference and Placebo in relation to the global assessment of local tolerability on the application site

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Giordan, Study Director — Fidia Farmaceutici s.p.a.
Locations (16):
- Germany (2):
  - Praxis Dr. med. Helmut Pabst, Gilching
  - Praxis Dr. Jürgen Ulrich Schaale-Maas, Rheinbach
- Hungary (12):
  - Synexus Budapest DRC, Budapest
  - Magyar Honvédség, Egészségügyi Központ Baleseti Sebészeti Osztály, Budapest
  - Uzsoki utcai Kórház Ortopéd-traumatológiai Osztály, Budapest
  - Synexus Debrecen AS, Debrecen
  - Platán Egészségcentrum, Eger
  - Synexus Magyarország kft. Gyula DRS, Gyula
  - Shawfar-med Kft, Kalocsa
  - Jutrix Kft., Kecskemét
  - Bács-Kiskun Megyei Kórház Kiskunfélegyházi Városi Kórház és Rendelőintézet, Kiskunfélegyháza
  - G&V Pharma-Med Bt., Makó
  - Nagyatádi Kórház Reumatológiai Osztály, Nagyatád
  - Synexus Magyarország EÜ szolg Kft., Zalaegerszeg
- Italy (2):
  - Ambulatorio MMG dott. Paolo Picco, Sant'Olcese Chiesa, Genova
  - Ambulatorio MMG dott. Andrea Pedemonte, Genova

IPD SHARING:
Plan to Share IPD: No